CLINICAL TRIAL: NCT00940693
Title: Pilot Study of the Efficacy of Duloxetine in Treating Adults With Attention Deficit Hyperactivity Disorder: a Randomized, Controlled Trial.
Brief Title: Pilot Study of Duloxetine in Adult Attention Deficit Hyperactivity Disorder(ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Smadar Valérie Tourjman, Centre Hospitalier Universitaire de Montréal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09.008
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-12

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Disorder with Hyperactivity; Duloxetine; Adult; ADDH; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- duloxetine (Active Comparator)
  Interventions: Drug: duloxetine
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: duloxetine — 60 mg capsule once per day for 6 weeks
  Other Names: cymbalta
  Arms: duloxetine
Drug: placebo — one capsule of placebo taken one a day for 6 weeks
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether duloxetine is an effective treatment of attention deficit disorder in adults.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ADHD of at least moderate intensity
* Able to give consent
* Able to swallow capsules

Exclusion Criteria:

* Allergic or do not tolerate duloxetine
* Under psychotherapy for ADHD
* Taking a medication that interacts with duloxetine, including all psychotropic medication
* Treated with medication for ADHD
* Unstable medical condition
* Severe renal insufficiency
* Liver insufficiency
* Substance/alcool abuse or dependency in the last 6 months
* Pregnancy, nursing or inadequate contraceptive methods
* Suicide or homicide risk
* Organic brain syndrome
* Any diagnosis of lifetime bipolar disorder or psychotic disorder, and any actual diagnosis of anxious disorder or major depressive disorder

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Impact of duloxetine on the Conners' Adult attention-Deficit/Hyperactivity Disorder Rating Scale-Observer Report:Screening Version (CAARS-O:SV) in adult ADHD subjects. | baseline and week 6

SECONDARY OUTCOMES:
Impact of duloxetine on the Clinical Global Impression Scale in ADHD adults | baseline and week 6
Impact of duloxetine on the Conners' Adult attention-Deficit/Hyperactivity Disorder Rating Scale-Self Report : Long Version(44) (CAARS-S:L), in adult ADHD subjects. | baseline and week 6
Impact of duloxetine on anxious and depressive symptoms in adult ADHD subjects. | baseline and week 6
Impact of duloxetine on Quality of life in adults with ADHD | baseline and week 6
Impact of duloxetine on executive functions and cognitive performances in adults with ADHD | baseline and week 6

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Tourjman, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier Universitaire de Montréal: Hôpital Notre-Dame, Montreal, Quebec, Canada

REFERENCES:
- [Background] Tourjman SV, Bilodeau M. Improvement with duloxetine in an adult ADHD patient. J Atten Disord. 2009 Jul;13(1):95-6. doi: 10.1177/1087054708326109. Epub 2009 Apr 9. PMID 19359667